CLINICAL TRIAL: NCT02069678
Title: Serum Hepatitis B Surface Antigen Levels to Guide the Stopping of Entecavir in HBeAg-negative Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Henry LY Chan, Professor, Chinese University of Hong Kong
Other Study IDs: Stop Nuc
Record Dates: First submitted 2014-01-28; First posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This will be a multi-center study in Hong Kong. This is a retrospective-prospective study in HBeAg-negative chronic hepatitis B patients. HBeAg-negative patients on entecavir followed up in the liver clinics will be identified from the existing database. All patients had HBV DNA testing every 6 months as a clinic routine. Serum HBsAg levels will be tested in the residual serum samples at the pre-treatment and last follow-up visits. Eligible patients will be discussed on the plan of stopping entecavir therapy. All patients will have written informed consent before recruited into this study. All patients will be followed up for 12 months after stopping entecavir treatment. As entecavir is most commonly used antiviral drug in Hong Kong and in the Western countries, the investigators aim to investigate and validate the use of serum HBsAg quantification to guide the timing of stopping entecavir in HBeAg-negative patients. The results of this study will provide scientific evidence on the use of this new serum marker to predict sustained remission after stopping entecavir. In the long-run, it can improve patient compliance, reduce the need of long-term antiviral and reduce the drug cost in the management of HBeAg-negative chronic hepatitis B.

All patients will stop entecavir according to the Asian Pacific guideline with written informed consent and close subsequent monitoring. In the protocol, there is a safety net for re-treatment. There will not be any invasive procedure. There is no major ethical issue.

DETAILED DESCRIPTION:
Chronic hepatitis B is the commonest cause of liver cirrhosis and hepatocellular carcinoma in Hong Kong. Approximately 50% of patients had negative hepatitis B e antigen (HBeAg), which indicates an escape of host immune clearance by the host. Oral antiviral drugs are very effective in suppressing viral replication and inducing biochemical remission [1]. However, the timing to stop oral antiviral agents is controversial. Hepatitis B surface antigen (HBsAg) seroclearance has been recommended as the best time for drug cessation for HBeAg-negative patients [2,3], but its occurrence is very uncommon especially among Asian patients. The Asian Pacific guideline recommended stopping treatment when serum HBV DNA became undetectable for three times within 12 months [4], but approximately 50% of patients will experience virologic relapse post-treatment [5,6].

HBsAg quantification has been shown to correlate with the concentration of covalently closed circular DNA in the liver [7]. In a Hong Kong study among 53 HBeAg-negative patients who stopped lamivudine, HBsAg ≤ 100 IU/ml and/or reduction of > 1 log at the end of treatment could predict sustained response up to 5 years post-treatment [8]. In other words, it is probable that patients who have a lower serum HBsAg level, which may reflect a lower concentration of virus inside the liver, have a lower risk of viral relapse after stopping antiviral therapy.

ELIGIBILITY:
Inclusion Criteria:

1. HBeAg-negative patients on entecavir monotherapy for at least 24 months
2. Undetectable HBV DNA by PCR-based assay on 3 separate occasions 6 months apart (as per Asian Pacific guideline in 2008).
3. Normal ALT levels according to the local laboratory reference value on 2 separate occasions 6 months apart

Exclusion Criteria:

1. Patients previously or currently on interferon therapy
2. Patients who have experienced another antiviral agent besides entecavir
3. Patients with hepatitis C virus infection as indicated by a positive anti-HCV serology test
4. Patients with Child's B liver cirrhosis, cirrhotic complications or hepatocellular carcinoma
5. Patients with organ transplantation
6. Serious medical illnesses or malignancy
7. Age < 18 years or > 65 years
8. No patient consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HBeAg-negative patients on entecavir followed up in the liver clinics will be identified from the existing database. All patients had HBV DNA testing every 6 months as a clinic routine. Serum HBsAg levels will be tested in the residual serum samples at the pre-treatment and last follow-up visits. Eligible patients will be discussed on the plan of stopping entecavir therapy. All patients will have written informed consent before recruited into this study. All patients will be followed up for 12 months after stopping entecavir treatment.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
sustained response, defined as HBV DNA persistently ≤ 200 IU/ml | 12 months after stopping Entecavir

SECONDARY OUTCOMES:
HBsAg < 1000 IU/ml and 100 IU/ml | 12 months post-treatment
HBV DNA < 200 IU/ml and 20 IU/ml | 12 months post-treatment
virological relapse | 5 years post-treastment
HBsAg clearance | 5 years post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng Suen Man Shook Hepatitis Center, Institute of Digestive Disease, The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Lai CL, Shouval D, Lok AS, Chang TT, Cheinquer H, Goodman Z, DeHertogh D, Wilber R, Zink RC, Cross A, Colonno R, Fernandes L; BEHoLD AI463027 Study Group. Entecavir versus lamivudine for patients with HBeAg-negative chronic hepatitis B. N Engl J Med. 2006 Mar 9;354(10):1011-20. doi: 10.1056/NEJMoa051287. PMID 16525138
- [Background] Lok AS, McMahon BJ. Chronic hepatitis B. Hepatology. 2007 Feb;45(2):507-39. doi: 10.1002/hep.21513. No abstract available. PMID 17256718
- [Background] European Association For The Study Of The Liver. EASL Clinical Practice Guidelines: management of chronic hepatitis B. J Hepatol. 2009 Feb;50(2):227-42. doi: 10.1016/j.jhep.2008.10.001. Epub 2008 Oct 29. No abstract available. PMID 19054588
- [Background] Liaw YF, Leung N, Kao JH, Piratvisuth T, Gane E, Han KH, Guan R, Lau GK, Locarnini S; Chronic Hepatitis B Guideline Working Party of the Asian-Pacific Association for the Study of the Liver. Asian-Pacific consensus statement on the management of chronic hepatitis B: a 2008 update. Hepatol Int. 2008 Sep;2(3):263-83. doi: 10.1007/s12072-008-9080-3. Epub 2008 May 10. PMID 19669255
- [Background] Chan HL, Wang H, Niu J, Chim AM, Sung JJ. Two-year lamivudine treatment for hepatitis B e antigen-negative chronic hepatitis B: a double-blind, placebo-controlled trial. Antivir Ther. 2007;12(3):345-53. PMID 17591024
- [Background] Chan HL, Wong VW, Tse AM, Tse CH, Chim AM, Chan HY, Wong GL, Sung JJ. Serum hepatitis B surface antigen quantitation can reflect hepatitis B virus in the liver and predict treatment response. Clin Gastroenterol Hepatol. 2007 Dec;5(12):1462-8. doi: 10.1016/j.cgh.2007.09.005. PMID 18054753
- [Background] Chan HL, Wong GL, Chim AM, Chan HY, Chu SH, Wong VW. Prediction of off-treatment response to lamivudine by serum hepatitis B surface antigen quantification in hepatitis B e antigen-negative patients. Antivir Ther. 2011;16(8):1249-57. doi: 10.3851/IMP1921. PMID 22155906